CLINICAL TRIAL: NCT04455126
Title: Preservative-free Tafluprost Eye Drops in Newly Diagnosed Patients With Glaucoma: A Prospective Clinical Study
Brief Title: Preservative-free Tafluprost Eye Drops in Newly Diagnosed Patients With Glaucoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Amir abou Samra, Prof., Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0105556
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: This was an open-label, non-randomized clinical study that aimed to assess the ocular signs and symptoms in 60 eyes of 30 newly diagnosed Egyptian glaucoma patients receiving preservative-free tafluprost eye drops.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preservative-free tafluprost (Experimental): This was an open-label, non-randomized clinical study that aimed to assess the ocular signs and symptoms in 60 eyes of 30 newly diagnosed Egyptian glaucoma patients receiving preservative-free tafluprost eye drops
  Interventions: Drug: Preservative-free tafluprost eye drops

INTERVENTIONS:
Drug: Preservative-free tafluprost eye drops — This was an open-label, non-randomized clinical study that aimed to assess the ocular signs and symptoms in 60 eyes of 30 newly diagnosed Egyptian glaucoma patients receiving preservative-free tafluprost eye drops

SUMMARY:
Glaucoma encompasses a collective group of optic neuropathies characterized by progressive degeneration of retinal ganglion cells and their axons, resulting in cupping, a distinctive appearance of the optic disc, and a pattern of visual loss

DETAILED DESCRIPTION:
Saflutan® is the first preservative-free prostaglandin analog introduced to the Egyptian market. It contains the PG analog tafluprost. Better tolerability, higher adherence to treatment and improvement of patients' quality of life are associated with using preservative-free eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females, newly diagnosed with glaucoma, naïve to glaucoma medications and surgery, able to read, comprehend, and complete the Ocular Surface Disease Index (OSDI) questionnaire, and able to provide informed consent form.

Exclusion Criteria:

* Unable to provide informed consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | 12 weeks
  Intraocular pressure (IOP)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Doheim, Principal Investigator — Alexandria Faculty of Medicine
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No